CLINICAL TRIAL: NCT04160026
Title: Acceptability and Feasibility of IPTp With Dihydroartemisinin-piperaquine With or Without Azithromycin to Prevent Malaria, Sexually Transmitted and Reproductive Tract Infections in HIV-uninfected Pregnant Women (IMPROVE) in Kenya.
Brief Title: Acceptability and Feasibility in the Context of the IMPROVE Trial in Kenya
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Liverpool School of Tropical Medicine (Other)
Collaborators: Kenya Medical Research Institute (Other); Kamuzu University of Health Sciences (Other); National Institute for Medical Research, Tanzania (Other Government); London School of Hygiene and Tropical Medicine (Other); University of Bergen (Other); Kilimanjaro Christian Medical Centre, Tanzania (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 18-073
Record Dates: First submitted 2019-11-07; First posted 2019-11-12 (Actual); Last update posted 2021-04-15 (Actual); Status verified 2021-04

CONDITIONS: Malaria in Pregnancy; Adherence, Treatment
MeSH Terms: conditions — Treatment Adherence and Compliance | interventions — fanasil, pyrimethamine drug combination

STUDY DESIGN:
Intervention Model Description: The feasibility study is cluster randomised, where a health facility is a cluster.
  The acceptability studies are nested within the feasibility study and the IMPROVE clinical trial.
Masking Description: The feasibility study in the routine setting was not masked, this was a 3-arm study where interventions were delivered by ministry of health staff.
  The acceptability study was nested in the clinical trial which was a 3-arm placebo controlled multicentre trial (see NCT02909712) .
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- IPTp-SP (Active Comparator): Arm 1. Standard single-day stat course of quality-assured SP (Fansidar ®) of 3 tablets (500 mg of sulphadoxine and 25 mg of pyrimethamine). SP given monthly
  Interventions: Drug: Monthly intermittent preventive treatment with sulfadoxine-pyrimethamine
- IPTp-DP (Experimental): Arm 2. Standard 3-day course of 3 to 5 tablets (40/320mg) of DP per day based on bodyweight (Eurartesim®, AlfaSigma, Italy). DP given monthly
  Interventions: Drug: Monthly intermittent preventive treatment with dihydroartemisnin-piperaquine
- IPTp-DP Plus (Experimental): Arm 3. Standard 3-day course of 3 to 5 tablets (40/320mg) of DP per day based on bodyweight (Eurartesim®, AlfaSigma, Italy) plus targeted information for health providers.
  Interventions: Drug: Monthly intermittent preventive treatment with dihydroartemisnin-piperaquine with targeted information transfer

INTERVENTIONS:
Drug: Monthly intermittent preventive treatment with dihydroartemisnin-piperaquine — Feasibility study to assess adherence among health providers in antenatal clinics delivering the study interventions in a routine setting and uptake and adherence among pregnant women.
  Other Names: Dihydroartemisnin- piperaquine -Eurartesim®
  Arms: IPTp-DP
Drug: Monthly intermittent preventive treatment with sulfadoxine-pyrimethamine — Feasibility study to assess adherence among health providers in antenatal clinics delivering the study interventions in a routine setting and uptake and adherence among pregnant women.
  Other Names: Sulfadoxine-Pyrimethamine; Control Arm
  Arms: IPTp-SP
Drug: Monthly intermittent preventive treatment with dihydroartemisnin-piperaquine with targeted information transfer — Feasibility study to assess adherence to guidelines among health providers in antenatal clinics delivering the study interventions in a routine setting and uptake and adherence among pregnant women.
  Other Names: Dihydroartemisnin- piperaquine -Eurartesim®; DP Plus
  Arms: IPTp-DP Plus

SUMMARY:
This multi-centre study will compare the acceptability, feasibility, cost and incremental cost-effectiveness of intermittent preventive treatment (IPTp) with dihydroartemisinin-piperaquine (DP) with or without azithromycin to the current strategy of IPTp with sulphadoxine-pyrimethamine (SP) to prevent malaria, sexually transmitted and reproductive tract infections in HIV-uninfected pregnant women (IMPROVE).

DETAILED DESCRIPTION:
Primary objectives:

1. To assess the acceptability, costs and incremental cost-effectiveness of IPTp-DP, with or without AZ, compared to current policy of IPTp-SP in HIV-uninfected pregnant women.
2. To assess the feasibility of delivering IPTp-DP with or without a targeted information transfer intervention among HIV-uninfected pregnant women attending ANC in the routine health system i.e. non-trial settings.

Acceptability, costs and incremental cost-effectiveness will be assessed in the context of the IMPROVE clinical trial in Kenya, Malawi and Tanzania (see NCT02909712).

We will also conduct an 'implementation feasibility' study in the routine setting in adjacent sites to the IMPROVE trial site in Kenya (only), using a 3-arm cluster randomized design to assess systems effectiveness, implementation strength, scalability, and identify potential operational hurdles for scale up. Ministry of health nurses providing routine ANC services will be trained to provide IPTp-DP or given refresher training for current policy (IPTp-SP). The interventions will be implemented for a period of 10 months. Approximately 5-6 months after the start of implementation, delivery effectiveness will be assessed through exit interviews with pregnant women leaving ANC clinics. Women who receive the correct doses of the interventions will be followed up at home 4-5 days after their clinic visit (i.e. no more than 2 days after their 3-day regimen finished) and interviewed about adherence, including pill counts. The quantitative study will be supplemented by a qualitative study to explain the quantitative outcomes and to assess perceptions of scalability of the interventions tested.

Feasibility study Interventions:

Monthly IPTp regimens: Arm 1. Standard single-day stat course of quality-assured SP; Arm 2. Standard 3-day course of 3 to 5 tablets (40/320mg) of DP per day based on bodyweight (Eurartesim®, AlfaSigma, Italy); Arm 3. Same as 2, with additional job aids and IEC materials.

Outcome Measures

Feasibility study:

Primary Outcome - Adherence assessed through home visits: Proportion of pregnant women attending ANC who receive the first dose of IPTp by DOT and the correct number of tablets for subsequent doses (IPTp-DP) visited at home and who have verified they completed the treatment. Where IPTp-SP is given by DOT this is assumed as 100% adherence and that the correct dosage is given.

Secondary outcome - Delivery effectiveness assessed by exit interviews with pregnant women leaving ANC: Proportion of pregnant women attending ANC for their first and second visit in their second or third trimester who receive an appropriate dose with each drug/drug combination. For the IPTp-DP arm, women will be asked whether the first dose was given by DOT and the correct number of tablets for subsequent doses available on exit. For IPTp-SP the full dose should be given by DOT.

Sample sizes:

Feasibility exit interviews (delivery rate): 1,485 pregnant women Feasibility home visits (adherence rate): 744 pregnant women sampled from women enrolled in exit interviews Acceptability among pregnant women: approx. 90 Acceptability among health providers: approx.90

ELIGIBILITY:
Inclusion Criteria:

* Kenya Government owned health facilities, Level 3 or 4 health facilities
* Pregnant women attending ANC through non-trial health facilities for a scheduled antenatal care visit in the second or third trimester who receive one of the three study interventions depending on which arm is allocated to that health facility

Exclusion Criteria:

* Mission or private health facilities, Kenya government owned Level 2 or level 5 health facilities, health facilities included in the trial
* Pregnant women accessing private health facilities
* Health facilities, or pregnant women, involved in other malaria or HIV in pregnancy intervention trials or studies.
* Pregnant women in the first trimester, or pregnant women for who their last visit was less than one month ago

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 1600 (Actual)
Dates: Start 2019-11-11 (Actual); Primary Completion 2020-07-31 (Actual); Study Completion 2020-07-31 (Actual)

PRIMARY OUTCOMES:
Adherence in pregnant women | Assessed 6-10 months after implementation commences
  Proportion of pregnant women attending ANC who receive the drug course correctly and who have verified they completed the treatment at home during a home visit.

SECONDARY OUTCOMES:
Effectiveness of service delivery | Assessed 6-10 months after implementation commences
  Proportion of pregnant women attending ANC for their first and second visit in their second or third trimester who receive the drug course correctly on exit from ANC. For IPTp-SP the full dose should be given by DOT.

CONTACTS AND LOCATIONS:
Overall Officials: Jenny Hill, PhD, Principal Investigator — Liverpool School of Tropical Medicine
Locations (1):
- Kenya Medical Research Institute, Kisumu, Kenya

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Barsosio HC, Webster J, Omiti F, K'Oloo A, Odero IA, Ojuok MA, Odiwa D, Omondi B, Okello E, Dodd J, Taegtmeyer M, Kuile FOT, Lesosky M, Kariuki S, Hill J. Delivery effectiveness of and adherence to intermittent preventive treatment for malaria in pregnancy with dihydroartemisinin-piperaquine with or without targeted information transfer or sulfadoxine-pyrimethamine in western Kenya: a three-armed, pragmatic, open-label, cluster-randomised trial. Lancet Glob Health. 2024 Oct;12(10):e1660-e1672. doi: 10.1016/S2214-109X(24)00261-4. PMID 39304238